CLINICAL TRIAL: NCT02297854
Title: Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-sequence, Cross Over, Single Dose, Oral Bioequivalence Study of Valganciclovir Hydrochloride Tablets 450 mg Under Fasting Condition
Brief Title: Bioavailability Study of Valganciclovir Hydrochloride Tablets 450 mg Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 569-10
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2011-09

CONDITIONS: Healthy
MeSH Terms: interventions — Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valganciclovir Hydrochloride Tablets 450 mg (Experimental): Valganciclovir Hydrochloride Tablets 450 mg of Dr. Reddys Laboratories Limited
  Interventions: Drug: Valganciclovir Hydrochloride
- Valcyte (Active Comparator): Valcyte® 450 mg tablets of Genentech USA Inc., San Francisco
  Interventions: Drug: Valganciclovir Hydrochloride

INTERVENTIONS:
Drug: Valganciclovir Hydrochloride — Valganciclovir Hydrochloride Tablets 450 mg
  Other Names: Valcyte

SUMMARY:
This study is to assess the Valganciclovir Hydrochloride Tablets 450 mg of Dr. Reddy's Laboratories Limited, India and Valcyte® (Valganciclovir HCl) tablets 450 mg of Genentech USA Inc., Group of Roche, South San Francisco in healthy, adult, human subjects under Fasting conditions.

DETAILED DESCRIPTION:
Open label, balanced, randomized, two-treatment, two-period, two-sequence, cross over, single dose, oral bioequivalence study of Valganciclovir Hydrochloride Tablets 450 mg under Fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, human volunteers between 18 to 55 years of age (both inclusive) living in and around Ahmedabad city or western part of India.
* Having a Body Mass Index (BMI) between 18.5-24.9 (both inclusive), calculated as weight in kg / height in meter2.
* Not having any significant disease in medical history or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations, 12- lead ECG and X-ray chest (postero-anterior view) recordings.
* Able to understand and comply with the study procedures, in the opinion of the principal investigator.
* Able to give voluntary written informed consent for participation in the trial.

In case of Male subjects:

* Willing to practice an acceptable barrier contraception method of birth control for the entire duration of the study and at least for 90 days after the last dose administration, and in case of an accidental pregnancy of their spouse should be willing to abort the pregnancy. Or
* Surgically sterile who have undergone vasectomy.

In case of female subjects:

* Surgically sterilized (Bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) at least 6 months prior to study participation; Or
* If of child bearing potential is willing to use a suitable and effective double barrier contraceptive method or intra uterine device of birth control or abstinence for the entire during of the study and at least 90 days after the last study drug administration and in case of an accidental pregnancy should be willing to abort the pregnancy. Or
* Postmenopausal women: Women who are postmenopausal for at least 1 year having Follicle stimulating Hormone (FSH) level and serum estradiol level (without hormone replacement therapy) within specified limit suggestive of menopausal state, having normal bilateral mammogram and normal ultrasound abdomen and pelvis. And
* Pregnancy test must be negative. No female volunteers were enrolled in the trial.

Exclusion Criteria :

The exclusion criteria as per the protocol were as follows:

* Known hypersensitivity or idiosyncratic reaction to Valganciclovir and/or ganciclovir or any of the excipients or any related drug.
* History or presence of any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
* Ingestion of a medicine at any time within 14 days before dosing in Period I. In any such case subject selection will be at the discretion of the Principal Investigator.
* Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAID induced urticaria.
* A recent history of harmful use of alcohol(less than 2 years), i.e. alcohol consumption of more than 14 standard drinks per week for men and more than 7 standard drinks per week for women (A standard drink is defined as 360 ml of beer or 150 ml of wine or 45 ml of 40% distilled spirits, such as rum, whisky, brandy etc) or consumption of alcohol or alcoholic products within 48 hours prior to receiving study medicine.
* Smokers, who smoke 10 or more than 10 cigarettes / day or inability to abstain from smoking during the study
* The presence of clinically significant abnormal laboratory values during screening.
* Use of any recreational drugs or history of drug addiction or testing positive in prestudy drug scans.
* History or presence of psychiatric disorders.
* A history of difficulty in donating blood.
* Donation of blood (1 unit or 350 mL) or receipt of an investigational medicinal product or participation in a drug research study within a period of 90 days prior to the first dose of study medication. Elimination half-life of the study drug should be taken into consideration for inclusion of the subject in the study. Note: In case the blood loss is ≤ 200 mL; subject may be dosed 60 days after blood donation or last sample of the previous study.
* A positive hepatitis screen including hepatitis B surface antigen and HCV antibodies.
* A positive test result for HIV antibody.
* An unusual diet, for whatever reason (e.g. low-sodium), for four weeks prior to receiving the study medicine. In any such case subject selection will be at the discretion of the Principal Investigator.
* Consumption of grape fruit or grape fruit products within 48 hours prior to dosing.
* Nursing mothers (females). No female volunteers were enrolled in the trial.Nursing mothers (females).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | 0.00 and at 0.167, 0.333, 0.50, 0.667, 0.833, 1.00, 1.25, 1.50, 1.75, 2.00, 2.333, 2.667, 3.00, 3.333, 3.667, 4.00, 6.00, 8.00, 10.00, 12.00, 16.00 and 24.00 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Aplesh kumar Patel, MD, Principal Investigator — Lambda Therapeutic Research Ltd.
Locations (1):
- Lambda Therapeutic Research Ltd, Ahmedabad, Gujarat, India